CLINICAL TRIAL: NCT04085133
Title: Prevalence and Burden of Bronchiectasis in Tuberculous Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Shaddad, DR.Ahmad Shaddad, Assiut University
Other Study IDs: 12345817
Record Dates: First submitted 2019-05-28; First posted 2019-09-11 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Tuberculoses
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Sputum by gene xpert
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gene Xpert Chest x ray and MSCT chest — Sputum sample for T.B will be done using gene expert device and chest xray and high resolution ct to evaluate bronchectasis

SUMMARY:
Bronchiectasis was described in the early 19th century by Laennec. Bronchiectasis is a chronic condition characterized by permanent and irreversible dilatation of the bronchial airways and impairment of mucociliary transport mechanism due to repeated infection and inflammation leading to colonization of organism and pooling of the mucus in the bronchial tree

DETAILED DESCRIPTION:
Bronchiectasis was described in the early 19th century by Laennec. Bronchiectasis is a chronic condition characterized by permanent and irreversible dilatation of the bronchial airways and impairment of mucociliary transport mechanism due to repeated infection and inflammation leading to colonization of organism and pooling of the mucus in the bronchial tree.

The prevalence of bronchiectasis is age-related and occurs in every age group and in the pre-antibiotic era . it most often began in childhood. Recent evidence shows that bronchiectasis disproportionately affects women and older individuals and will be contributing to increase in healthcare burden.[3] International data show an increase in the prevalence of bronchiectasis over recent years.

ELIGIBILITY:
Inclusion Criteria:

* 1-patients were diagnosed to have tuberculosis by sputum culture and gene x pert.

  2-patients were diagnosed to have bronchiectasis after lab and radiological examination as well as clinical score.

  3- patients diagnosed as bronchiectasis after history of tuberculosis or anti Tuberculosis treatment with positive or negative tuberculous culture in the time of research.

Exclusion Criteria:

* 1-patients presented with other Pulmonary diseases. 2-Chronic liver and renal disease . 3- Lung cancer and tumors. 4- patients were previously diagnosed as bronchiectasis .

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Any tuberculosis patients admited to assuit university hospital and assuit chest hospital
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
To study prevalence of bronchiectasis in TB patients by case per year. | One year
  How many patients of TB will be diagnosed as abronchiectasis

SECONDARY OUTCOMES:
To evaluate the burden of bronchiectasis in TB patients | one year
  by frequency of need for hospital admission per year, need for outpatient clinical visits per month and frequency of need for antimicrobial therapy other than anti-tuberculous treatment per month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut unviresty, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided